CLINICAL TRIAL: NCT07019025
Title: Development and Implementation of a Structured Therapeutic Education Program on the Use of Mobile Applications for People With Diabetes Mellitus.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitales Universitarios Virgen del Rocío (Other)
Responsible Party: Principal Investigator, Pilar Santa Cruz Álvarez, MSc, Advanced Diabetes Nurse, Hospitales Universitarios Virgen del Rocío
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MPSA-CB-2024
Record Dates: First submitted 2024-10-03; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; nurses
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bolus calculation (Experimental): The intervention will consist of a structured therapeutic education program led and taught by nurses based on the use of mobile applications to manage glycemic control, reinforce self-efficacy and improve knowledge of the disease. It will be carried out over 3 face-to-face group sessions of a maximum of 5 consecutive people in the CDT, another with the same characteristics after 90 days and an individual telematic session after 6 months. The hospitalization or internalization of the person was established as criteria to interrupt or modify the intervention. To improve compliance with the protocol and intervention, periodic meetings will be agreed upon with the nurses in charge of education.
  Interventions: Other: Therapeutic patient education on the use of a insulin bolus calculator app

INTERVENTIONS:
Other: Therapeutic patient education on the use of a insulin bolus calculator app — Therapeutic patient education on the use of a insulin bolus calculator app

SUMMARY:
Introduction:

Diabetes mellitus (DM) is a group of disorders characterized by chronic hyperglycemia due to issues with insulin production or function. Globally, the incidence is about 15 cases per 100,000 people, with a prevalence of 9.5%. In Spain, the highest prevalence rates are in the Canary Islands, Murcia, and Castilla y León. DM management includes a balanced diet, exercise, medication, and therapeutic education. Nurse-led programs improve patient outcomes, and mobile apps like Social Diabetes and MySugar help calculate insulin dosages based on diet and other factors.

Methodology:

The study will take place at the Hospital Universitario Virgen del Rocío in Seville, Spain. Participants will be selected based on eligibility criteria, including being over 18, having diabetes under basal-bolus treatment, and being able to use a mobile phone. Exclusion criteria include cognitive impairment and severe illnesses.

The intervention includes a structured education program led by nurses using mobile apps, with 3 group sessions and one individual session at 6 months. The primary outcome is glycemic control, and secondary outcomes include self-efficacy and knowledge levels. The study requires 52 participants, with data collected by nurse educators and analyzed using SPSS. Ethics approval and informed consent will be obtained. The authors declare no conflicts of interest.

DETAILED DESCRIPTION:
Introduction:

Diabetes mellitus (DM) comprises a group of metabolic disorders characterized by chronic hyperglycemia due to abnormalities in insulin production or function. Globally, the incidence is approximately 15 cases per 100,000 people, with a prevalence of 9.5%. In Spain, there is significant prevalence among adults and children, with the highest rates observed in the Canary Islands, Murcia, and Castilla y León.

DM management focuses on a balanced diet, physical exercise, pharmacological treatment, and therapeutic education to reduce morbidity and mortality. Nurse-led therapeutic education programs have proven effective in improving self-control and health outcomes in DM patients. Mobile applications like Social Diabetes and MySugar have gained relevance, facilitating the calculation of necessary insulin boluses according to carbohydrate intake and other parameters.

Objective:

To analyze the effect of a structured therapeutic education program on glycemic control, self-efficacy, and knowledge in people with diabetes mellitus under basal-bolus treatment. A specific objective is to design and implement a structured therapeutic education program for adjusting insulin boluses relative to diet using mobile apps. The study will be conducted as a longitudinal inferential research with random assignment.

Methodology:

The study will be conducted at the Diagnostic and Treatment Center of Hospital Universitario Virgen del Rocío (HUVR) in Seville, Spain. Participants will be selected following nurse assessment of eligibility criteria. Inclusion criteria include being over 18 years old with diabetes mellitus under basal-bolus treatment and owning and being able to use a mobile phone. Exclusion criteria include cognitive impairment, having acute or chronic exacerbated illnesses at recruitment, and lack of temporal and geographical availability.

The intervention will consist of a structured therapeutic education program led by nurses using mobile applications. It will be conducted in 3 group sessions and one individual telematic session at 6 months. The primary outcome will be glycemic control measured through the ambulatory glucose profile (AGP). Secondary outcomes will measure self-efficacy and knowledge levels.

The required sample size was calculated to be 52 participants. Data collection will be carried out by nurse educators and analyzed using SPSS version 29. Approval from the Biomedical Research Ethics Committee of Andalusia will be sought, and informed consent will be obtained from participants.

The authors declare no conflicts of interest.

ELIGIBILITY:
The inclusion criteria will be to be over 18 years old with Diabetes Mellitus in bolus/basal treatment, to have and know how to use one's own mobile phone. The exclusion criteria will consist of cognitive impairment, having acute or worsening chronic diseases at the time of recruitment and lack of temporal and geographical availability.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Control glucémico | March 2025
  The main outcome will be glycemic control through the values collected in the ambulatory glucose profile (AGP) report (time in range, time below range, time above range, coefficient of variability, average glucose, management indicator of glucose)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen del Rocío, Seville, Sevilla, Spain